CLINICAL TRIAL: NCT06686992
Title: The Effect of Distraction Method on Children's Pain and Fear Levels During Vaccine Administration: a Randomized Controlled Trial
Brief Title: The Effect of Distraction Method on Children's Pain and Fear Levels During Vaccine Administration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, ARZU SARIALİOĞLU, Associate professor, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: B.30.2.ATA.0.01.00/134
Record Dates: First submitted 2024-11-12; First posted 2024-11-13 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2024-11

CONDITIONS: Vaccination
Keywords: pain; fear; vaccine; nursing; distraction; child
MeSH Terms: conditions — Pain | interventions — Vaccination

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- distraction (Experimental): The researcher will fill in the questionnaire and scales 5 minutes before the vaccination. During the procedure, the child will be played with roll-and-draw. The scales will be filled in again 5 minutes after the procedure. It will take an average of 5-10 minutes to fill out the forms.
  Interventions: Behavioral: Vaccination
- control (No Intervention): Questionnaires and scales will be filled out by the researcher 5 minutes before vaccination. Only routine applications will be made. The scales will be filled again 5 minutes after vaccination.

INTERVENTIONS:
Behavioral: Vaccination — The researcher will fill in the questionnaire and scales 5 minutes before the vaccination. During the procedure, the child will be played with roll-and-draw. The scales will be filled in again 5 minutes after the procedure. It will take an average of 5-10 minutes to fill out the forms.
  Arms: distraction

SUMMARY:
The study will be conducted to examine the effect of distraction method on children's pain and fear levels during vaccine administration. The research will be conducted in a randomized controlled experimental design in Family Health Centers in a province in eastern Turkey between November and December 2024. The population of the study will consist of children who come to the Family Health Center to receive the 4-year-old vaccine. The study will be completed with 50 intervention and 50 control groups, totaling 100 children. Child Diagnostic Information Form, Wong-Baker Facial Expression Rating Scale and Child Fear Scale will be used to collect the data. Children in the intervention group will play the roll and draw game before and during vaccination. Children in the control group will receive routine vaccination. Research ethical principles will be followed.

DETAILED DESCRIPTION:
The research will be conducted in a randomized controlled experimental design in Family Health Centers in a province in eastern Turkey between November and December 2024. The population of the study will consist of children who come to the Family Health Center to receive the 4-year-old vaccine. The study will be completed with 50 intervention and 50 control groups, totaling 100 children. Child Diagnostic Information Form, Wong-Baker Facial Expression Rating Scale and Child Fear Scale will be used to collect the data. Children in the intervention group will play the roll and draw game before and during vaccination. Children in the control group will receive routine vaccination. Research ethical principles will be followed.

Round and Draw game: The game designed by the researcher will be used as the intervention tool in the study. The game is played by creating a face picture by drawing the corresponding sections with the help of a dice consisting of 6x5 sections. With the game, it is planned to minimize pain and fear in children during vaccination. Care will be taken to ensure that the materials to be used are appropriate for the developmental level of the children, easy to clean and do not develop any allergies in children.

Data Collection The researcher will be present in the centers where the study will be conducted for 1 day to examine the ergonomic structure of the pediatric family health centers before starting to collect the data of the play group and control group children. The children and their parents will be given preliminary information about the research (the purpose of the research, why the research is being conducted, the use of the roll-and-draw game in relieving the child's pain and fear, etc.), and after obtaining verbal consent from the children and written consent from the parents, the data of the research will be obtained by face-to-face interview method with the children who agree to participate in the research.

Control Group: The questionnaires and scales will be filled in by the researcher 5 minutes before the vaccination process. Only routine 4-year-old vaccines will be administered. The scales will be filled out again 5 minutes after the procedure. It will take an average of 5-10 minutes to fill out the forms.

Interventıon Group: The questionnaire and scales will be filled out by the researcher 5 minutes before vaccination. During the procedure, the child will be played with roll-and-draw. The scales will be filled in again 5 minutes after the procedure. It will take an average of 5-10 minutes to fill out the forms.

ELIGIBILITY:
Inclusion Criteria:

* Being 4 years old
* Not having a disability related to developmental areas
* The mother or father should be with the child during the procedure

Exclusion Criteria:

* being older or younger than 4 years old
* having a chronic disease
* lack of willingness to work

Ages: 4 Years to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-03-12 (Actual)

PRIMARY OUTCOMES:
Wong-Baker Facial Expression Rating Scale (WB-FRAS) | 1 months
  This scale is used to diagnose pain in children aged 3-18 years. In this scale, there are six faces representing increasing pain intensity from zero to five from left to right. The leftmost face has a smiling expression, indicating a pain-free state, while the rightmost face has a crying expression, corresponding to the most severe pain. The child is instructed to choose the face that best expresses their own emotions. Six facial expressions are scored from left to right from 0 to 5 points (0 points= very happy/no pain, 5 points= most severe pain). As the score obtained from the scale increases, pain tolerance decreases and as the score decreases, tolerance increases.
Child Fear Scale | 1 months
  The Child Fear Scale was developed in 2011 to measure fear in children undergoing painful medical procedures. The Child Fear Scale is a 0-4 scale with five faces ranging from neutral (0 = no concern at all) to fearful (4 = severe concern).

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University Nursing of Faculty, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.